CLINICAL TRIAL: NCT04803994
Title: The ABC-HCC Trial: A Phase IIIb, Randomized, Multicenter, Open-label Trial of Atezolizumab Plus Bevacizumab Versus Transarterial Chemoembolization (TACE) in Intermediate-stage HepatoCellular Carcinoma
Brief Title: The ABC-HCC Trial: Atezolizumab Plus Bevacizumab vs. Transarterial Chemoembolization (TACE) in Intermediate-stage HepatoCellular Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ABC-HCC; 2020-004210-35 (EudraCT Number); 2024-512953-26-00 (EU CTIS Number)
Record Dates: First submitted 2021-03-15; First posted 2021-03-18 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma; HCC; intermediate stage; atezolizumab; bevacizumab; TACE
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Clinical trial with two study arms:
  Experimental arm A: 50% of the patients will receive a combination therapy (systemic) of the monoclonal antibodies atezolizumab and bevacizumab.
  Control arm B: 50% of the patients will receive TACE therapy (locoregional).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systemic therapy with atezolizumab + bevacizumab (Experimental): Patients receive atezolizumab 1200 mg flat dose plus bevacizumab 15 mg/kg given intravenously every 3 weeks until failure of strategy, participant request, or withdrawal of consent for a maximum of up to 24 months.
  The discontinuation of one of the study drugs for toxicity reasons does not qualify as failure of treatment strategy as long as the other drug can be continued according to protocol.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab
- Locoregional therapy with TACE (Active Comparator): Patients will receive initial TACE and - if required to achieve or improve an objective response - a second TACE after 8 weeks (±7 days window). Thereafter, additional TACE can be applied on demand until failure of strategy, participant request, or withdrawal of consent for a maximum of up to 24 months.
  TACE must be discontinued in cases of technical difficulties making additional TACE impossible.
  Only conventional TACE (cTACE) and drug-eluting bead TACE (DEB-TACE) approaches are accepted as TACE therapy. However, consistency in the TACE procedure and the use of the chemotherapeutic agent has to be maintained for each individual patient.
  Interventions: Procedure: TACE

INTERVENTIONS:
Drug: Atezolizumab — 1200 mg atezolizumab intravenously Q3W (max 32 cycles, up to 24 months)
  Other Names: Tecentriq
  Arms: Systemic therapy with atezolizumab + bevacizumab
Drug: Bevacizumab — 15 mg/kg intravenously Q3W (max 32 cycles, up to 24 months)
  Other Names: Avastin
  Arms: Systemic therapy with atezolizumab + bevacizumab
Procedure: TACE — Locoregional therapy will be performed as a standard-of-care procedure
  Other Names: transarterial chemoembolization
  Arms: Locoregional therapy with TACE

SUMMARY:
The ABC-HCC trial is a Phase IIIb, randomised, multicenter, open-label study designed to evaluate the safety and efficacy of atezolizumab plus bevacizumab versus TACE in patients with intermediate-stage HCC. Approximately 434 patients in two arms of treatment will be enrolled.

DETAILED DESCRIPTION:
The main purpose of this phase IIIb study is to test the efficacy and safety of atezolizumab in combination with bevacizumab compared to TACE in patients with intermediate stage liver cancer.

Primary efficacy objective is to assess the efficacy of atezolizumab in combination with bevacizumab compared to TACE in patients with intermediate stage liver cancer.

The secondary efficacy objective is to further characterize the responses obtained with the respective therapeutic strategy and to assess the impact of each therapeutic strategy on liver function over time.

Furthermore the objective is to evaluate the safety and tolerability of each therapeutic strategy and their respective impact on Quality of Life and to identify prognostic and predictive angiogenic and immune related biomarkers (tissue and circulating) for study endpoints.

This is a Phase IIIb, randomised, multicenter, open-label study. Approximately 434 patients suffering from intermediate-stage hepatocellular carcinoma will be enrolled in this trial. Patients will be recruited from up to 60 sites in 10 different countries.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form available
2. Patients* ≥ 18 years of age at time of signing Informed Consent Form
3. Confirmed hepatocellular carcinoma diagnosis based on histopathological findings from tumor tissue or typical diagnostic imaging on dynamic CT or MRI according to AASLD criteria.
4. Intermediate stage HCC as defined by the following criteria:

   * Disease not amenable to curative surgery, liver transplantation or curative ablation BUT disease amenable to TACE at enrollment as judged by the investigator.
   * No massive multinodular pattern preventing adequate TACE
   * No tumor of a diffuse infiltrative HCC type (hypovascular infiltrative tumors with ill-defined borders)
   * Patent portal vein flow
   * No main portal vein invasion/thrombosis on baseline/eligibility imaging. Patients with minimal invasion, (Vp1 and Vp2) may be eligible if no exclusion criteria are violated.
   * No extrahepatic disease Note: Patients with HCC beyond Milan criteria who enter a downstaging protocol may be recruited into the trial if they do not present any exclusion criteria.
5. Patients with recurrence after resection/ablation or after previous TACE are eligible, if they - according to the investigator - have an indication for (additional) TACE
6. Child-Pugh score class A or B7 without ascites requiring more than 100 mg of spironolactone/day (see exclusion criteria) at enrollment.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 at enrollment.
8. Adequate organ and bone marrow function
9. Life expectancy of ≥ 3 months
10. The following laboratory values obtained less than or equal to 7 days prior to randomization.

    * Total bilirubin ≤ 3.0 x the upper limit of normal (ULN)
    * Urine dipstick for proteinuria ≤ 2+ (within 7 days prior to randomization) Patients discovered to have ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate < 1 g of protein in 24 hours
    * The following other laboratory values measured within 7 days prior to randomization are either normal or if abnormal do not represent a medical contraindication for TACE and atezolizumab/bevacizumab as judged by the investigator: Platelet count, hemoglobin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), serum creatinine, INR or aPTT, alkaline phosphatase, neutrophil count (ANC), and serum albumin.
11. Negative serum pregnancy test done lesser than or equal to 7 days prior to randomization, for females of childbearing potential only.
12. No presence of untreated or incompletely treated varices with bleeding or high-risk for bleeding: Availability of esophagogastroduodenoscopy (not older than 6 months) in which all size of varices (small to large) had been assessed and varices were treated per local standard of care prior to randomization.
13. Absence of other severe comorbidities
14. Resolution of any acute, clinically significant treatment-related adverse events from prior therapy/procedure to Grade ≤ 1 prior to randomization, with the exception of alopecia.
15. For patients with active hepatitis B virus (HBV):

    * HBV DNA ≤ 2000 IU/mL obtained within 28 days prior to randomization, AND
    * Anti-HBV treatment (per local standard of care; e.g., entecavir) for a minimum of 14 days prior to randomization and willingness to continue treatment for the length of the study.
16. For patients with active hepatitis C virus (HCV):

    * Patients positive for hepatitis C virus (HCV) antibody are eligible, also if polymerase chain reaction testing is positive for HCV ribonucleic acid (RNA).
    * However, anti-viral therapy against HCV is only allowed prior to trial but not during the trial.
    * For HBV and HCV co-infection refer to exclusion criterion # 11.
17. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for at least 5 months after the last dose of atezolizumab, 6 months after the last dose of bevacizumab, or 1 month after the last TACE procedure.

    * A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).
    * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
    * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
18. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below:

    * With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for 6 months after the last dose of bevacizumab or 1 month after the last TACE procedure. Men must refrain from donating sperm during this same period.
    * With pregnant female partners, men must remain abstinent or use a condom during the treatment period and for 6 months after the last dose of bevacizumab or 1 month after the last TACE procedure to avoid exposing the embryo.
    * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

      * There are no data that indicate special gender distribution. Therefore, patients will be enrolled in the study gender-independently.

Exclusion Criteria:

1. 1. Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC (only if proven by biopsy).
2. Previous treatment with atezolizumab or bevacizumab.
3. Previous treatment with a programmed death 1 (PD1), programmed death-ligand (PD-L1), or cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) inhibitors, or any form of cancer immunotherapy for HCC.
4. Clinically meaningful ascites, defined as ascites requiring non-pharmacologic intervention (e.g. paracentesis) to maintain symptomatic control.

   • Patients with ascites requiring pharmacologic intervention (e.g. diuretics) and stable for ≥ 2 months on low doses of diuretics (spironolactone 100 mg/d or equivalent) for ascites are eligible. Of note, diuretics for other indications such as congestive heart failure are not considered in this regard.
5. Major surgical procedure, open biopsy, or significant traumatic injury ≤ 28 days prior to randomization or anticipation of need for major surgical procedure during the course of the study or non-recovery from side effects of any such procedure.
6. Significant cardiovascular disease, such as cardiac disease (New York Heart Association Class II or greater), myocardial infarction or cerebrovascular accident within 3 months prior to randomization, as well as unstable arrhythmias (note: beta blockers or digoxin are permitted), unstable angina, new-onset angina (begun within the last 3 months).
7. Uncontrolled hypertension defined by a systolic blood pressure (BP) ≥ 150 mmHg or diastolic blood pressure (BP) ≥ 100 mmHg, with or without antihypertensive medication. Prior history of hypertensive crisis or hypertensive encephalopathy. Patients with initial blood pressure (BP) elevations are eligible if initiation or adjustment of antihypertensive medication lowers pressure to meet entry criteria.
8. Current or recent (within 10 days prior to study treatment start) use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic purpose (prophylactic anticoagulation permitted, e.g. new oral anticoagulants [apixaban, dabigatran, rivaroxaban], LMW heparin, ASA up to 300 mg/qd).
9. Arterial or venous thrombotic or embolic events such as cerebro-vascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism ≤6 months prior to randomization.
10. With regards to eligibility for adequate TACE, patients presenting with either of the following conditions are excluded:

    * Past history of bilioenteric anastomosis or biliary procedure (e.g., endoscopic papillotomy or biliary stenting) or patients with aerobilia
    * Central biliary obstruction (right or left intrahepatic duct, common hepatic duct, common bile duct)
    * Celiac occlusion
11. Any ongoing infection > grade 2 NCI-CTCAE version 5.0. Note on HIV, HBV, and HCV infection: also consider inclusion criteria #s 15, 16, and exclusion criterion # 18. Patients with co-infection for HBV and HCV are excluded, unless tested negative for HCV RNA by PCR.
12. Patients with seizure disorder requiring medication.
13. Prior allogeneic bone marrow transplantation or prior solid organ transplantation.
14. Evidence or history of bleeding diathesis or any hemorrhage or bleeding event > CTCAE grade 3 within 4 weeks prior to randomization.
15. Non-healing wound, ulcer, or bone fracture.
16. Renal failure requiring hemo- or peritoneal dialysis.
17. Known hypersensitivity to any of the study drugs, study drug classes, or excipients in the formulation including a history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion protein; known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab or bevacizumab formulation.
18. Positive test for human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS), with the following exception: patients with a positive HIV test at screening are eligible, provided they are stable on anti-retroviral therapy, have a CD4 count > 200 cells/µL, and have an undetectable viral load.
19. Active tuberculosis
20. Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
21. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, idiopathic pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest computed tomography (CT) scan Note: History of radiation pneumonitis within the radiation field (fibrosis) is permitted.
22. Persistent proteinuria of CTCAE Grade 3 or higher (> 3.5 g/24 hrs, measured by urine protein: creatinine ratio on a random urine sample).
23. Pregnant or nursing women
24. Comorbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens.
25. Active or history of autoimmune disease including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener's granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.

    Note: History of autoimmune-mediated hypothyroidism on a stable dose of thyroid replacement hormone, or controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible based on consultation with the sponsor's medical monitor. Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:
    * Rash must cover < 10% of body surface area
    * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
    * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months.
26. Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-α agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

    * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study.
    * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
27. Use of any herbal remedies known to interfere with the liver or other major organ functions. Patients must notify the investigator of all herbal remedies used during the study.
28. Administration of a live, attenuated vaccine within four weeks prior to start of enrollment, or anticipation that such a live attenuated vaccine will be required during the study or within 5 months after the last dose of atezolizumab, 6 months after the last dose of bevacizumab, or 1 month after the last TACE procedure.
29. History of malignancy other than HCC within 3 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g. 5-year OS rate > 90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer. Other similar cases can be considered after discussion with lead investigators and sponsor.
30. Receipt of an investigational drug within 28 days prior to initiation of study drug
31. Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent or patients with substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Time to failure of treatment strategy | 48 months - assessed every 8 weeks (±7days)
  The primary endpoint is defined as the time from randomization until death or need for a further therapeutic option, defined for each arm as follows:
  * Arm A: Time from randomization until the failure of strategy does not allow for further treatment with atezolizumab + bevacizumab; or death, whichever comes first.
  * Arm B: Time from randomization until the failure of strategy does not allow for further TACE therapy; or death, whichever comes first.
  Failure of strategy (in brief): failure of strategy is reached in case of progressive disease accompanied by any of the following: loss of clinical benefit, unacceptable toxicity, liver function deterioration, therapy not further applicable for other reasons.

SECONDARY OUTCOMES:
Overall survival (OS) | 48 months
  Time from the date of randomization until the date of death due to any cause. A subject who has not died will be censored at last known date alive.
Overall Survival Rate at 24 months (OS@24) | 24 months
  The proportion of patients assigned to a treatment arm known to be alive at 24 months after randomization.
Objective Response Rate (ORR) | 48 months
  The proportion of patients assigned to a treatment arm with a confirmed best response of Complete Response (CR) or Partial Response (PR). Response will be assessed according to HCC mRECIST.
Time to Progression (TTP) | 48 months
  Time from the date of randomization until the date of first objective disease progression. Subjects who have not progressed will be censored at the last evaluable tumor assessment date prior to subsequent anti-cancer therapy. Subjects who die without experiencing a progress first will be censored on their date of death.
Time to loss of systemic treatment options (TTSYS) | 24 months
  Time from the date of randomization until the date the patient reaches a state of being unfit for any subsequent systemic treatment option (BSC as only option left) or the date of death whichever occurs first. Subjects who end systemic treatment at their own request will be censored at the day of end of systemic treatment. Subjects who are lost to follow-up will be censored at the date last known to be systemically treated.
Progression free survival (PFS) | 48 months
  Time from the date of randomization until the date of first objective disease progression or death. Subjects who did not progress or die will be censored at the last evaluable tumor assessment date prior to subsequent anti-cancer therapy.
Duration of Treatment | 24 months
  From start of treatment to permanent discontinuation of the treatment arms A and B.
Duration of Response (DOR) | 48 months
  Time from initial response to progressive disease or death in patients in treatment arms A and B with a confirmed best response of Complete Response (CR) or Partial Response (PR) according to HCC mRECIST. Subjects who did not progress or die will be censored at the last evaluable tumor assessment date prior to subsequent anti-cancer therapy.
Time to deterioration of liver function | 48 months
  Time from the date of randomization until liver function deterioration is registered according to definition given for failure of strategy. Only patients experiencing a deterioration of liver function are included into this analysis
Treatment-related and -unrelated toxicities (AEs, SAEs) according to NCI CTCAE v5.0 | 48 months
  Summary of adverse events by treatment arm and CTCAE (version 5.0) grade and frequency of clinically significant abnormal laboratory parameters.
QoL (EORTC QLQ-C30 and HCC18 sub-questionnaire) | 48 months
  QoL mean values and response as well as time to symptom deterioration (TTSD) defined as the time interval between randomization and the first decrease by ≥ 10-points. All randomly assigned patients with a baseline and at least one post-baseline assessment will be included in TTSD analyses. Patients without observed deterioration will be censored at the time of their last QoL assessment.

OTHER OUTCOMES:
Exploratory endpoint - Correlation of biomarkers for study endpoints | 48 months
  Tissue, blood and stool samples will be collected to identify prognostic and predictive angiogenic and immune related biomarkers (tissue and circulating) for study endpoints.
Exploratory endpoint - PD-L1 expression | 48 months
  PD-L1 expression will be analyzed by immunohistochemistry on available FFPE tissue samples

CONTACTS AND LOCATIONS:
Overall Officials: Salah Eddin Al-Batran, Prof. Dr., Study Director — Institut für Klinische Krebsforschung IKF GmbH, Frankfurt, Germany; Peter Galle, Prof. Dr., Principal Investigator — Universitätsmedizin Mainz, Germany; Jordi Bruix, Prof. Dr., Principal Investigator — Barcelona Clinic Liver Cancer, Universitat de Barcelona, Spain
Locations (72):
- Austria (6):
  - LKH - Univ. Klinikum Graz, Graz
  - Medzinische Universität Innsbruck, Innsbruck
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Ordensklinikum Linz, Linz
  - Universitätsklinikum St. Pölten, Sankt Pölten
  - Medizinische Universität Wien, Vienna
- France (10):
  - Institut Sainte-Catherine, Avignon
  - Hôpital Jean-Verdier Avicenne, Bobigny
  - CHU Bordeaux, Bordeaux
  - CHU Clermont-Ferrand CHU Estaing, Clermont-Ferrand
  - Beaujon Hospital, Clichy
  - CHU Grenoble, Grenoble
  - Croix-Rousse Hopital, Lyon
  - Saint Joseph Hopital - Marseille, Marseille
  - Hôpital Universitaire Pitié Salpêtrière, Paris
  - Centre Hépato-biliaire Paul Brousse, Villejuif
- Germany (26):
  - University Hospital RWTH Aachen, Aachen
  - Klinikum St. Marien Amberg, Amberg
  - Vivantes Klinikum Neukölln, Berlin
  - Universitätsklinikum Bochum, Bochum
  - Uniklinik Köln, Cologne
  - Universitätsklinikum Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Erlangen, Erlangen
  - Klinikum Esslingen, Esslingen am Neckar
  - Universitätsklinikum Frankfurt, Frankfurt
  - Krankenhaus Nordwest, Frankfurt am Main
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsmedizin Göttingen, Göttingen
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum Konstanz, Konstanz
  - Krankenhaus Maria-Hilf Krefeld, Krefeld
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Universitätsmedizin Mainz, Mainz
  - Universitätsklinikum Mannheim, Mannheim
  - Universitätsklinikum Marburg, Marburg
  - Klinikum rechts der Isar München, München
  - Klinikum Mutterhaus Trier, Trier
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
  - Uniklinik Ulm, Ulm
  - St. Josefs Hospital Wiesbaden, Wiesbaden
  - Universitätsklinikum Würzburg, Würzburg
- Italy (6):
  - Policlinico S. Orsola Bologna, Bologna
  - Instituto Tumori della Romagna IRST IRCCS, Meldola
  - Policlinico di Milano, Milan
  - Instituto di Tumori, Milan
  - Università di Pisa (UNIPI), Pisa
  - AOUI Verona, Verona
- Japan (9):
  - Hokkaido University Hospital, Hokkaido
  - Kobe University Hospital, Kobe
  - Kumamoto University Hospital, Kumamoto
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Nagasaki University Hospital, Nagasaki
  - Kindai University Hospital, Osaka
  - Saitama Medical University Hospital, Saitama
  - Fujita Health University Hospital, Toyoake
  - Yamaguchi University Hospital, Ube
- Spain (15):
  - Hospital Universitario de Alicante, Alicante
  - Hospital Infanta Cristina, Badajoz
  - Hospital Germans Trias I Pujol, Badalona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Barcelona Clinic Liver Cancer, Universitat de Bracelona, Barcelona
  - Hospital Puerta del Mar, Cadiz
  - Hospital de Jaen, Jaén
  - Hospital Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Fundación Jimenez Diaz, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Hospital de Alcorcón, Madrid
  - Hospital de Málaga, Málaga
  - Hospital Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.